CLINICAL TRIAL: NCT07371078
Title: Patient Satisfaction With Conventional, Additive and Subtractive Occlusal Splints for TMDs: A Clinical Randomized Trial
Brief Title: Conventional, Additive and Subtractive Occlusal Splints for TMDs
Acronym: TMD - TMJ - DD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mai Ahmed Haggag, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A010012024RP
Record Dates: First submitted 2026-01-03; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: TMD; Disc Displacement
Keywords: TMD; DDWR; CAD/CAM; 3D-printed; Occlusal Splint; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Splint (Experimental)
  Interventions: Device: Conventional Stabilizing Splint
- Milled Splint (Experimental)
  Interventions: Device: Milled Stabilizing Splint
- 3D Printed Splint (Experimental)
  Interventions: Device: 3D Printed Stabilizing Splint

INTERVENTIONS:
Device: Conventional Stabilizing Splint — Manual Manufacturing
  Arms: Conventional Splint
Device: Milled Stabilizing Splint — Subtractive Manufacturing
  Arms: Milled Splint
Device: 3D Printed Stabilizing Splint — Additive Manufacturing
  Arms: 3D Printed Splint

SUMMARY:
This study is aiming to clinically compare between occlusal splints produced by conventional, subtractive and additive techniques in regard to patient satisfaction.

DETAILED DESCRIPTION:
The development of a digital (CAD/CAM) technology incorporating three-dimensional (3D) printing and milling enabled the use of different materials and manufacturing techniques. However, it should be noted that most of the evidence is based on in vitro studies with different methodologies, limiting their validity in daily practice. To the authors knowledge, limited data in the literature clinically evaluated occlusal splints produced by conventional, subtractive and additive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of pain in the orofacial region (either arthrogenous and/or myogenous TMD) in the last 3 months.
* Patients never underwent any type of treatment for TMD's.
* Patients should have at least six natural teeth in each quadrant.

Exclusion Criteria:

* Any systemic condition associated with widespread pain (e.g., fibromyalgia).
* Medical history of current drug addiction.
* Patients with psychiatric disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Overall Patient Satisfaction | 6 months
  Using PSPSQ Questionnaire [The patient satisfaction questionnaire comprised three questions assessed using a 10-point Likert scale (1=extremely dissatisfied, 2=very dissatisfied, 3=dissatisfied, 4=slightly dissatisfied, 5=neutral, 6=slightly satisfied, 7=satisfied, 8=very satisfied, 9=extremely satisfied and 10=perfect/strongly satisfied)]
  * Scott AA, Hatch JP, Rugh JD, et al: Psychosocial predictors of satisfaction among orthognathic surgery patients. Int J Adult Orthodon Orthognath Surg 15:7, 2000
  * J. C. Posnick and J. Wallace, "Complex Orthognathic Surgery: Assessment of Patient Satisfaction," Journal of Oral and Maxillofacial Surgery 66, no. 5 (2008): 934-942.

SECONDARY OUTCOMES:
Time of adjustment | Baseline (At the time of occlusal splint delivery)
  Time of adjustment was measured in minutes
  - Algabr, R.S., Alqutaibi, A.Y., Elkadem, A.H., Maher, E.A., & Kaddah, A.F. (2017). Patient's satisfaction and muscles activity after management of temporomandibular disorders patients using computer-aided design/computer-aided manufacturing versus conventional occlusal splints (randomized clinical trial).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.researchgate.net/publication/313407164_Patient's_satisfaction_and_muscles_activity_after_management_of_temporomandibular_disorders_patients_using_computer-aided_designcomputer-aided_manufacturing_versus_conventional_occlusal_splints_random